CLINICAL TRIAL: NCT04782089
Title: A Phase II, Open, Single-center Study of PD-1 Antibody and PARP Inhibitor as Consolidation Treatment for Patients With Extensive Stage Small Cell Lung Cancer Who Have Not Progressed After First-line Treatment
Brief Title: Study of PD-1 Antibody and PARP Inhibitor in Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-2nd-IIT-SHR3162-APA
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Fluzoparib (Experimental)
  Interventions: Drug: Camrelizumab Anti-PD-1 antibody Fluzoparib PARP inhibitors

INTERVENTIONS:
Drug: Camrelizumab Anti-PD-1 antibody Fluzoparib PARP inhibitors — Camrelizumab+Fluzoparib：Q3W, Administration until disease progression or intolerable

SUMMARY:
This is a Phase II, Open, Single-center Study of Camrelizumab and Fluzoparib as Consolidation Treatment for Patients With Extensive stage small cell lung cancer Who Have Not Progressed after first-line treatment

ELIGIBILITY:
Inclusion Criteria:

1. All subjects were required to sign the informed consent before starting the study;
2. Histologically documented Extensive stage small cell lung cancer；
3. ECOG PS 0~1 ；
4. 18-75 years；
5. According to recist1.1, CR or PR was achieved after 4-6 cycles of first-line etoposide and platinum chemotherapy;
6. .Life expectancy ≥ 3 months；

Exclusion Criteria:

1. Recurrence or distant metastasis of localized small cell lung cancer after chemotherapy or concurrent chemoradiotherapy；
2. Active infection including tuberculosis, HIV, hepatitis B and C；
3. Interstitial pneumonia (ILD), drug-induced pneumonia, radiation-induced pneumonia requiring steroid therapy or active pneumonia with clinical symptoms, or other moderate to severe lung diseases that seriously affect lung function;
4. Severe infection existed, including but not limited to infection complications, bacteremia, severe pneumonia, etc;
5. Symptomatic brain metastasis and cancerous meningitis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 3 years
  To assess the efficacy of Camrelizumab and Fluzoparib combination therapy in terms of PFS